CLINICAL TRIAL: NCT01907607
Title: Efficacy and Safety of PD-0332991 in Patients With Advanced Gastrointestinal Stromal Tumors Refractory to Imatinib and Sunitinib: A Phase 2 Study
Brief Title: Efficacy and Safety of PD-0332991 in Advanced Gastrointestinal Stromal Tumors Refractory to Imatinib and Sunitinib
Acronym: CYCLIGIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB 2013-01
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2020-12

CONDITIONS: Advanced Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumor; PD-0332991; Efficacy; advanced; safety
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PD-0332991 (Experimental): Adult patients with Advanced Gastrointestinal Stromal Tumors Refractory to Imatinib and Sunitinib.
  PD-0332991 is formulated as gelatin capsules of 100 mg and 25 mg respectively.
  Interventions: Drug: PD 0332991

INTERVENTIONS:
Drug: PD 0332991 — PD-0332991 was administrated orally, formulated as gelatin capsules of 100 mg and 25 mg respectively.
  PD-0332991 was dosed on a flat scale of 125 mg (1 capsule x 100 mg/day, 1 capsule x25 mg/day) will be administrated orally o.d on a 21 days on / 7 days off dosing schedule. One cycle is considered to consist of 4 weeks of PD-0332991 administration.
  Patients should be instructed to administrate PD-0332991 with a sufficient amount of water at least 1 hour prior to a meal or at least 2 hours following a meal and to swallow the required number of capsules at approximately the same time on each day.

SUMMARY:
The treatment of advanced GIST patients is based on imatinib followed with sunitinib in case of resistance/intolerance. However, the median progression-free survival (PFS) on sunitinib is frequently short, and after failure with both imatinib and sunitinib, treatment remains controversial.

Previous studies on GISTs have linked 9p21 alterations to tumor progression (El-Rifai et al. 2000; Kim et al., 2000; Schneider-Stock et al., 2003; Schneider-Stock et al., 2005; Romeo et al. 2009; Haller et al., 2008) but the driver gene was not positively identified (CDKN2A, CDKN2B, or MTAP) (Astolfi et al., 2010; Belinsky et al., 2009; Perrone et al., 2005; Assamaki et al. 2007; Huang et al., 2009). A recent study has shown that homozygous 9p21 deletions target CDKN2A and more specifically p16INK4a 4. Most of the CINSARC genes are known to be under the transcriptional control of E2F. RB1 sequesters E2F, which is released from the complex upon RB1 phosphorylation by CDK4. CDK4 is, in turn, inhibited by p16INK4a. Hence, we hypothesize that alteration of the restriction point via deletion of p16INK4a (and more rarely of RB1: 20% of cases) gene in GISTs is likely to be a causative event that leads to the overexpression of CINSARC genes, which in turn induce chromosome instability and ultimately metastasis. Low p16INK4a expression was associated with response to PD-0332991 in several in vitro tumor model(Konecny et al. 2011; Katsumi et al. 2011; Finn et al. 2009). Considering our molecular data, we believed that PD-0332991 warrants clinical investigation in advanced gastrointestinal stromal tumors with alteration of p16INK4a. This alteration is detectable by comparative genomic hybridization which is a technique highly manageable in the context of routine clinical care and clinical trial.

Main objective was to assess the antitumor activity of PD-0332991 in terms of non-progression at 16 weeks (after centralized review) in patients with documented disease progression while on therapy with imatinib and sunitinib for unresectable and/or metastatic GIST.

DETAILED DESCRIPTION:
Medical Conditions : Adult patients with Advanced Gastrointestinal Stromal Tumors Refractory to Imatinib and Sunitinib

Study design : Exploratory, one-arm, multicenter, phase II clinical trial based on two-stage Simon's design

Main objective : To assess the antitumor activity of PD-0332991 in terms of non-progression at 16 weeks (after centralized review) in patients with documented disease progression while on therapy with imatinib and sunitinib for unresectable and/or metastatic GIST.

Secondary objectives

* To assess the antitumor activity of PD-0332991 in terms of :

  * Objective response rate (ORR) (as per RECIST v1.1 criteria)
  * Progression-free survival (PFS) (as per RECIST v1.1 criteria)
  * Overall survival
* To assess the safety of PD-0332991

Study drug formulation: PD-0332991 is formulated as gelatin capsules of 100 mg and 25 mg respectively. PD-0332991 was administrated orally. PD-0332991 dosed on a flat scale of 125 mg. PD-0332991 was administrated on a 21 days on / 7 days off dosing schedule. One cycle was considered to consist of 4 weeks of PD-0332991 administration.Patients were treated with PD-0332991 until progression of disease, unacceptable toxicity, death or discontinuation for any other reason.

Tumor assessment and response assessed according to RECIST v1.1, with same type of exam in regard of baseline.

All potential sites of tumor lesions (target and non-target lesions) assessed using MRI or CT Scan with IV contrast of the Thorax Abdomen and Pelvis using a 5mm slice thickness with a contiguous reconstruction algorithm (a PET scan is not acceptable for radiological evaluation).

Evaluation were assessed:

* at baseline within 21 days before the first dose of PD-0332991
* at D(28) of Cycle 1, at D(28) of Cycle 2 then every 8 weeks until month six and then every 12 weeks until disease progression or starting other treatment.

Response regarding the first endpoint was assessed by central radiology review. Whenever the criteria of response are met (Complete Response (CR) or Partial Response (PR)), the appropriate imaging tests were repeated at least four weeks later in order to confirm the response.

The decision regarding patient management remained with the local investigator.

optionnal: Fresh tumor biopsies FFPE (Formalin-Fixed Paraffin-Embedded) at screening and at Day 21 of Cycle 1 are encouraged to be collected. Once collected, the samples may be profiled by IHC, and array gene expression analysis

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age
2. Histologically confirmed GIST of any anatomical location and confirmed by the RRePS Network ; positive immunohistochemical staining for c-KIT (CD117); or negative staining for KIT, but with either positive staining for DOG1 or an identified mutation of KIT or PDGFRA gene
3. CDKN2A gene deletion assessed by array-comparative genomic hybridization (array-CGH)
4. Unresectable and/or metastatic disease with documented progression according to modified RECIST criteria (see section 7.2.1.5 of protocol) after 1st line imatinib and 2nd line sunitinib. Progression on the last line of treatment should be confirmed by central review with two radiological assessments identical (CT scans or MRI) obtained at less from 4 months interval within the 24 months before inclusion.
5. At least one measurable GIST lesion according to RECIST (v1.1 Appendix 3). A previously irradiated lesion is eligible to be considered as a measurable lesion provided that there is objective evidence of progression of the lesion prior to starting PD-0332991.
6. A performance status of 0, 1 or 2 according to the Eastern Cooperative Oncology Group (ECOG) scale(Appendix 1)
7. Recovery from Grade 2 to 4 toxicity related to prior line of treatment assessed according to NCICTCAE v.4.0 (Appendix 2)
8. Adequate bone marrow function as shown by:

   Blood absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   1. Blood platelets ≥ 100 x 109/L
   2. Blood hemoglobin (Hgb) > 9 g/dL
9. Adequate liver function as shown by:

   c. Serum or plasma ALT and AST ≤ 3.0 x ULN (regardless of the presence or absence of metastases) d. Serum or plasma total bilirubin: ≤ 1.5 x ULN (excepted for patients with Gilbert's syndrome)
10. Adequate renal function as shown by serum creatinine ≤ 2 x ULN
11. Patients who give a written informed consent obtained according to French and European regulations.
12. Patients affiliated to the French Social Security

Exclusion Criteria:

1. RB1 gene deletion assessed by array-comparative genomic hybridization (array-CGH)
2. Patients who received anti-cancer drugs ≤ 5 days prior to starting PD-0332991
3. Patients who are treated or planned to be treated concomitantly with other cytotoxic or antineoplastic treatments, such as chemotherapy, immunotherapy, biological response modifiers, or radiotherapy
4. Patients with another primary malignancy within 2 years prior to starting the study drug, with the exception of adequately treated in-situ carcinoma of the uterine cervix, or completely excised (R0 resection) basal or squamous cell carcinoma of the skin
5. Patients with a corrected QT interval using Bazett's formula (QTcB) > 470 msec.
6. Current use or anticipated need for food or drugs that are known strong cytochrome P450 (CYP)3A4 inhibitors (i.e. grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, posaconazole, erythromycin, clarithromycin, tilithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, nefazodone, diltiazem, and delaviridine)
7. Patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PD-0332991 (e.g. severe ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or extensive (>1m) small bowel resection, inability to swallow oral medications). Prior partial gastrectomy is not an exclusion criterion.
8. Patients with prior complete gastrectomy
9. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism.
10. Patients with any clinically significant medical or surgical condition which, according to investigators' discretion, should preclude participation

    1. i.e. active or uncontrolled infection, uncontrolled diabetes, active or chronic liver disease (cirrhosis, chronic active hepatitis or chronic persistent hepatitis)
    2. hepatitis B or C virus carriers with normal liver function tests, can be included
11. Known diagnosis of human immunodeficiency virus (HIV) infection. HIV testing is not mandatory
12. Patients who are currently receiving anticoagulation treatment with therapeutic doses :

    1. of warfarin or equivalent anticoagulant (e.g. high dose aspirin or clopidogrel or other)
    2. or have an INR >1.5. Treatment with acetylsalicyclic acid 100 mg daily or low molecular weight heparin (LMWH) is allowed
13. Pregnant or breast-feeding women
14. Women of child-bearing potential not employing two effective methods of birth control. Effective contraception must be used throughout the trial and 24 weeks after the end of PD-0332991 (e.g. condom with spermicidal jelly, foam suppository or film; diaphragm with spermicide; male condom and diaphragm with spermicide, oral, implantable, or injectable contraceptives). Women of child-bearing potential defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e. who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 21 days prior to starting study drug.
15. Fertile males not willing to use contraception as stated above
16. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Italiano, MD/PhD, Principal Investigator — Institut Bergonié
Locations (9):
- France (9):
  - Institut Bergonié, Bordeaux, Gironde
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone - AP-HM, Marseille
  - Centre René Gauducheau, Nantes
  - Hôpital Saint-Antoine (AP-HP), Paris
  - CHU de REIMS - Hôpital Robert Debré, Reims
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toulmonde M, Blay JY, Bouche O, Mir O, Penel N, Isambert N, Duffaud F, Bompas E, Esnaud T, Boidot R, Geneste D, Ghiringhelli F, Lucchesi C, Bellera CA, Le Loarer F, Italiano A. Activity and Safety of Palbociclib in Patients with Advanced Gastrointestinal Stromal Tumors Refractory to Imatinib and Sunitinib: A Biomarker-driven Phase II Study. Clin Cancer Res. 2019 Aug 1;25(15):4611-4615. doi: 10.1158/1078-0432.CCR-18-3127. Epub 2019 Apr 12. PMID 30979737

RESULTS

PARTICIPANT FLOW:
Groups:
- PD-0332991: Adult patients with Advanced Gastrointestinal Stromal Tumors Refractory to Imatinib and Sunitinib.
  PD-0332991 is formulated as gelatin capsules of 100 mg and 25 mg respectively.
  PD-0332991 will be administrated orally, formulated as gelatin capsules of 100 mg and 25 mg respectively.: PD-0332991 dosed on a flat scale of 125 mg (1 capsule x 100 mg/day, 1 capsule x25 mg/day) will be administrated orally o.d on a 21 days on / 7 days off dosing schedule. One cycle is considered to consist of 4 weeks of PD-0332991 administration.
  Patients should be instructed to administrate PD-0332991 with a sufficient amount of water at least 1 hour prior to a meal or at least 2 hours following a meal and to swallow the required number of capsules at approximately the same time on each day.
Period: Overall Study
Arm/Group | PD-0332991
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PD-0332991
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 66 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non Progression at 4 Months
Description: Efficacy is assessed based on 4-month non progression. Non progression is defined as complete or partial response (CR, PR) or stable disease (SD), using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Non-progression rate will be calculated as the number of alive and progression free patients divided by the number of eligible and assessable patients for the efficacy analysis. Eligible and assessable populations are described in corresponding section of protocol. As recommended by RECIST v1.1, all claimed response will be centrally reviewed by an expert of the study. The results of the centralized radiological review will be used for the analysis of the primary endpoint.
Time Frame: 16 weeks after first administration of treatment
Population: Population evaluable for efficacy: All patients eligible and for whom the following conditions are satisfied:
  (i) Received at least one complete or two incomplete treatment cycles, (ii) At least one disease measurement recorded not less than four weeks after treatment onset.
Measure: Count of Participants; unit: Participants
Arm/Group | PD-0332991
Number analyzed (Participants) | 23
Participants | 3

2. Secondary Outcome: Number of Participants With Objective Response at 4 Months
Description: Objective response is defined as complete response (CR) or partial response (PR) according to RECIST v1.1 Efficacy is assessed based on objective response at 4-month. Objective response is defined as complete or partial response (CR, PR) using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Objective reponse will be calculated as the number of alive patients with objective reponse divided by the number of eligible and assessable patients for the efficacy analysis. Eligible and assessable populations are described in corresponding section of protocol. As recommended by RECIST v1.1, all claimed response will be centrally reviewed by an expert of the study. The results of the centralized radiological review will be used for the analysis.
Time Frame: 16 weeks after first administration of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PD-0332991
Number analyzed (Participants) | 23
Participants | 0

3. Secondary Outcome: Efficacy Assessment of PD-0332991 in Terms of Progression-free Survival Time
Description: Progression-free survival time is defined as the time from the first administration of treatment to progression (as per RECIST v1.1) or death of any cause, whichever occurs first.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: up to 18 months following first administration of treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PD-0332991
Number analyzed (Participants) | 23
Months | 1.74 [0.92 to 3.45]

4. Secondary Outcome: Efficacy Assessment of PD-0332991 in Terms of Overall Survival Time
Description: Overall survival is defined as the time from the first administration of treatment to death.
Time Frame: up to 24 months following first administration of treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PD-0332991
Number analyzed (Participants) | 23
months | 19.52 [10.94 to 22.80]

ADVERSE EVENTS:
Time Frame: up to 24 months following first administration of treatment
Arm/Group | PD-0332991
All-Cause Mortality (participants affected / at risk) | 3/29
Serious Adverse Events (participants affected / at risk) | 12/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD-0332991 (N=29)
Flu-like syndrom (General disorders) | 1 (1)
Left ilio femoral phebilits (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Neutropenia (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal insuficiency (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Hemoperitoneum (Gastrointestinal disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Urinary infection (Infections and infestations) | 1 (1)
Deterioration of renal function (Renal and urinary disorders) | 1 (1)
Bladder globe (Renal and urinary disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric pain (Gastrointestinal disorders) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Sudden death at home (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD-0332991 (N=29)
Anemia (Blood and lymphatic system disorders) | 17 (22)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 6 (7)
Stomach pain (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 4 (4)
Fatigue (General disorders) | 10 (11)
Fever (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 2 (2)
Pain (General disorders) | 3 (3)
General disorders and administration site conditions (General disorders) | 3 (3)
Creatinine increased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 12 (17)
Platelet count increased (Investigations) | 4 (4)
White blood cell decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 4 (4)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders - Other (Renal and urinary disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
other (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Phlebitis (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT01907607/Prot_SAP_000.pdf